CLINICAL TRIAL: NCT05097157
Title: Feasibility Study To Assess A Radiofrequency Microneedling Device For Electrocoagulation And Hemostasis Of Soft Tissues For Dermatologic Conditions
Brief Title: Study To Assess A Radiofrequency Microneedling Device For Dermatologic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN19-RF-MN-01
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Wrinkle; Fine Lines; Crepey Skin; Acne Scars; Acne; Enlarged Pores; Stretch Marks; Loose Skin
MeSH Terms: conditions — Acne Vulgaris; Striae Distensae; Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment with Device (Experimental): Subjects received up to 5 treatments with the device, spaced 4 weeks apart.
  Interventions: Device: Potenza

INTERVENTIONS:
Device: Potenza — Subjects are treated with the Potenza™ device if they present with conditions such as, but not limited to: wrinkles, fine lines, crepey skin, acne scars, active acne, enlarged pores, stretch marks, or loose skin on the face, neck and/or body.

SUMMARY:
Subjects are to be enrolled in this clinical study if they are 18 - 55 years old. Up to 120 subjects will be enrolled at multiple study centers. Subjects may receive up to 5 treatments for a wide array of dermatologic conditions in which electrocoagulation and hemostasis is a viable mechanism for means of improvement.

ELIGIBILITY:
Inclusion Criteria:

* A healthy, non-smoking male or female between the age of 18-55 years old.
* Fitzpatrick skin type I to VI.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months prior to entering this study.
* The subject has physical problems such as cardiovascular disorders.
* The subject has a pacemaker.
* The subject had previous use of gold thread skin rejuvenation.
* The subject has skin infections.
* The subject has any of the following conditions:

  * Diabetes
  * Epilepsy
  * Acute disease
  * Dermatitis
* Subjects with electronic implants such as cardiac defibrillator. It may interfere with operation of electronic implants or damage the implants, causing risks.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.; Sean Doherty, Principal Investigator — Cynosure, Inc.; Robert Weiss, Principal Investigator — Maryland Dermatology Laser, Skin, & Vein Institute, LLC; Emil Tanghetti, Principal Investigator — Center for Dermatology and Laser Surgery; David McDaniel, Principal Investigator — McDaniel Institute of Anti-Aging Research
Locations (4):
- United States (4):
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Maryland Dermatology Laser, Skin, & Vein Institute, LLC., Hunt Valley, Maryland
  - Cynosure, Westford, Massachusetts
  - McDaniel Institute of Anti-Aging Research, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Device
Started | 79
Completed | 56
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Device
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants] — One subject was 72 years old and was given permission to enroll in the study per the investigator's discretion.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 78
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 72
  Hispanic | 4
  Asian | 1
  African American | 1
  Algerian/French | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Measure Description: The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale used is cited in the reference section
  Participants
    Fitzpatrick Skin Type I | 0
    Fitzpatrick Skin Type II | 32
    Fitzpatrick Skin Type III | 43
    Fitzpatrick Skin Type IV | 3
    Fitzpatrick Skin Type V | 0
    Fitzpatrick Skin Type VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction
Description: Subjects were asked to grade their satisfaction with the results of the treatment as either extremely dissatisfied, dissatisfied, slightly dissatisfied, slightly satisfied, satisfied, or extremely satisfied.
Time Frame: 30 day follow up
Population: 6 subjects were considered complete but did not have satisfaction information from their 30 day follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Device
Number analyzed (Participants) | 50
Participants
  Extremely Satisfied | 7
  Satisfied | 21
  Slightly Satisfied | 15
  Slightly Dissatisfied | 4
  Dissatisfied | 2
  Extremely Dissatisfied | 1

2. Primary Outcome: Global Aesthetic Improvement Scale Assessment (GAIS) Assessment
Description: The Clinical Global Aesthetic Improvement Scale (CGAIS) ranging from "worse" to "very much improved" is be used to judge the improvement as seen by the treating Investigator. The Investigator compared the baseline (pre-treatment) photographs to the follow up photographs to determine if the follow up image looks worse, if there is no change, if there is improvement, if there is much improvement, or if there is very much improvement in the follow up image when compared to the baseline image.
Time Frame: 30 day follow up
Population: 12 subjects were considered complete but did not have satisfaction information from their 30 day follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Device
Number analyzed (Participants) | 44
Participants
  Very Much Improved | 1
  Much Improved | 8
  Improved | 27
  No Change | 8
  Worsened | 0

3. Primary Outcome: Subject Satisfaction
Description: as for outcome 1
Time Frame: 90 day follow up
Population: 40 subjects did not complete the 90 day follow up for the subject satisfaction However, subjects who completed at least their 30 day follow up were considered complete. 1 subject had 2 different treatment areas treated and had a satisfaction score taken for both treatment areas.
Measure: Number; unit: treatment areas
Units Other Than Participants: treatment areas
Arm/Group | Treatment With Device
Number analyzed (Participants) | 15
Number analyzed (treatment areas) | 16
treatment areas
  Extremely Satisfied | 4
  Satisfied | 5
  Slightly Satisfied | 5
  Slightly Dissatisfied | 1
  Dissatisfied | 0
  Extremely Dissatisfied | 1

4. Primary Outcome: Global Aesthetic Improvement Scale Assessment (GAIS) Assessment
Description: as for outcome 2
Time Frame: 90 day follow up
Population: 41 subjects did not complete the 90 day follow up for the CGAIS. However, subjects who completed at least their 30 day follow up were considered complete. 1 subject had 2 different treatment areas treated and had a CGAIS taken for both treatment areas.
Measure: Number; unit: treatment areas
Units Other Than Participants: Treatment areas
Arm/Group | Treatment With Device
Number analyzed (Participants) | 15
Number analyzed (Treatment areas) | 16
treatment areas
  Very Much Improved | 0
  Much Improved | 5
  Improved | 10
  No Change | 1
  Worsened | 0

ADVERSE EVENTS:
Time Frame: Subject data was collected throughout subject participation in the study, approximately 9 months.
Arm/Group | Treatment With Device
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 0/79
Other Adverse Events (participants affected / at risk) | 37/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Device (N=79)
erythema (Skin and subcutaneous tissue disorders) | 37
Edema (Skin and subcutaneous tissue disorders) | 37
Pinpoint bleeding (Skin and subcutaneous tissue disorders) | 33
Burning sensation (Skin and subcutaneous tissue disorders) | 13
Dryness (Skin and subcutaneous tissue disorders) | 13
Scabbing (Skin and subcutaneous tissue disorders) | 9
Skin Textural Irregularity (Skin and subcutaneous tissue disorders) | 9
Bruising (Skin and subcutaneous tissue disorders) | 6
Pain/tenderness (Skin and subcutaneous tissue disorders) | 6
Tightness (Skin and subcutaneous tissue disorders) | 5
Itching (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Breakout (Skin and subcutaneous tissue disorders) | 3
Streaking (Skin and subcutaneous tissue disorders) | 4
Pain (Skin and subcutaneous tissue disorders) | 3
Burn (Skin and subcutaneous tissue disorders) | 4
Stabbing sensastion post pinpoint bleeding (Skin and subcutaneous tissue disorders) | 1
Tearing (Eye disorders) | 1
Eye twitch (Eye disorders) | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Rash/skin irritation (Skin and subcutaneous tissue disorders) | 1
Histamine (General disorders) | 1
Blanching (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Sensitivity (Skin and subcutaneous tissue disorders) | 1
Pinpoint dots (Skin and subcutaneous tissue disorders) | 1
Tingling (Skin and subcutaneous tissue disorders) | 1
Pustule (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05097157/Prot_SAP_000.pdf